CLINICAL TRIAL: NCT01936233
Title: Liver Cancer Institiute ,Fudan University
Brief Title: Clinical Study of Antiviral and Aspirin Treatment in Liver Cancer After Radical Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zheng-Gang Ren, chief of departement, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC-ASPIRIN
Record Dates: First submitted 2013-09-02; First posted 2013-09-06 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2018-12

CONDITIONS: Hepatocellular Carcinoma; Recurrence
Keywords: Hepatocellular Carcinoma; Aspirin; antiviral treatment; recurrence free survival; radical therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Aspirin; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin AND Lamivudine (Experimental)
  Interventions: Drug: Aspirin; Drug: Lamivudine
- Lamivudine (Active Comparator)
  Interventions: Drug: Lamivudine

INTERVENTIONS:
Drug: Aspirin — Aspirin 0.1 QD po
  Arms: Aspirin AND Lamivudine
Drug: Lamivudine — LAminvudine 0.1 QD po

SUMMARY:
Evaluation the Treatment Outcome of Antiviral and Aspirin Treatment in Liver Cancer After Radical Surgery.

DETAILED DESCRIPTION:
The investigators conduct this clinical trial to evaluate the treatment outcome of Antiviral and Aspirin Treatment in Liver Cancer After Radical Surgery.The primary outcome is overall survival and objective response rate.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma confirmed with pathology or identified with radiological images with typical features
* Age ≥ 18 years and ≤ 75 years
* At least one tumor nodule with one uni-dimension of ≥ 2 cm
* Child-Pugh Class A or B
* HBV-DNA>10^4
* Total bilirubin ≤ 1.5 x upper limit of normal
* ALT and AST ≤ 2.0 x the upper limit of normal
* PT-INR<2.3,PTT < 1.5 x upper limit of normal
* Serum creatinine ≤ 1.5x upper limit of normal
* Peripheral white blood cell count of or more than 3×10(9)/L
* Peripheral platelet of or more than 50×10(9)/L
* Expected survival time not less than 3 months
* ECOG score 0-2

Exclusion Criteria:

* Tumor thrombi in main branch of portal vein
* Tumor involvement more than 70% of whole liver
* With extrahepatic metastasis
* Prior systemic chemotherapy or chemoembolization
* Congestive heart failure > NYHA class 2
* History of HIV infection
* Active clinically serious infections (> 2 NCI-CTC Version 3.0)
* Recurrence of HCC after liver transplantation
* Pregnant or breast-feeding
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in this study
* Known or suspected allergy to any agent given in association with this trial
* Patients unable to swallow oral medication
* Inclined to thrombosis
* Inclined to hemorrhage or active hemorrhage with 1 month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2013-08; Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
recurrence free survival | 36 months

SECONDARY OUTCOMES:
overall survival | 36 months
adverse events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhenggang Ren, Ph.D, Principal Investigator — Fudan University
Locations (1):
- Liver Cancer Institute, Shanghai, Shanghai Municipality, China